CLINICAL TRIAL: NCT00608764
Title: Genetic Epidemiology of Chronic Obstructive Pulmonary Disease (COPDGene)
Brief Title: Examining the Genetic Factors That May Cause Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPDGene
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Edwin K. Silverman, Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 1428; 75N92023D00011-0-7 (Other: NHLBI); U01HL089856 (NIH); U01HL089897 (NIH)
Record Dates: First submitted 2008-01-28; First posted 2008-02-06 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Emphysema; Chronic Bronchitis; Genetics; Association Studies; Computed Tomography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic DNA, RNA, serum, and plasma will be collected and stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- NHW COPD Participants: Non-Hispanic white participants with COPD
- NHW Control Group: Non-Hispanic white participants with normal spirometry (do not have COPD)
- AA COPD Participants: African-American participants with COPD
- AA Control Group: African-American participants with normal spirometry (do not have COPD)

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a long-term lung disease that is often caused by cigarette smoking. The purpose of this study is to evaluate whether certain genetic factors predispose some smokers to develop COPD more than others.

DETAILED DESCRIPTION:
COPD is a disease in which the lung airways are damaged and partly obstructed, making it difficult to breathe. Millions of people in the United States have COPD, and it is the third leading cause of death in the United States. Symptoms include coughing, excess mucus production, shortness of breath, wheezing, and chest tightness. Emphysema and long-term bronchitis are the two most common manifestations of the disease. The most common risk factor for developing COPD is cigarette smoking; however, only 15% to 20% of smokers develop COPD in their lifetimes. It is not known why some smokers develop COPD and some do not, but certain genetic factors, combined with exposure to cigarette smoke, may increase the likelihood of developing COPD. This study will analyze DNA from current and former cigarette smokers to identify genetic factors and markers that may indicate a predisposition to developing COPD.

This study will enroll African-American and white cigarette smokers and former cigarette smokers both with and without COPD. Participants will attend one study visit during which they will complete questionnaires about lung symptoms, breathing difficulties, medical and family history, and quality of life. They will also undergo blood collection, a physical exam, lung function testing, and a walking test to measure endurance. Participants will undergo a high resolution computed tomography (CT) chest scan and a medical record review. Study researchers will contact participants up to four times a year for 15 years to collect follow-up medical information. Five-year, ten-year, and fifteen-year follow-up visits including a similar study protocol as the baseline visit will be performed on all available subjects.

ELIGIBILITY:
Inclusion Criteria:

* At least 10 pack-years of cigarette smoking (although a of nonsmoking controls is also being enrolled)
* Self-designation of non-Hispanic white or African-American

Exclusion Criteria:

* Other lung diseases (except for asthma in participants with COPD)
* Pregnant
* Cancer (other than skin cancer) in the 5 years prior to study entry
* Received antibiotics for a COPD exacerbation in the 1 month prior to study entry
* First- or second-degree relative of a previously enrolled study participant

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Particpants with COPD will include outpatient clinic patients, patients in registries, previous study participants, and COPD Foundation volunteers.
  Participants without COPD will include spouses and friends of study participants with COPD and patients at primary care practices.
Sampling Method: Non-Probability Sample
Enrollment: 10718 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | Measured at baseline
Emphysema, as shown on chest CT scan | Measured at baseline
Airway wall thickness on chest CT scan | Measured at baseline
COPD status (COPD participants versus control group participants) | Measured at baseline

CONTACTS AND LOCATIONS:
Overall Officials: James D. Crapo, MD, Principal Investigator — National Jewish Health; Edwin K. Silverman, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Diego, San Diego, California
  - Los Angeles Biomedical Research Institute, Torrance, California
  - National Jewish Health, Denver, Colorado
  - Morehouse School of Medicine, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Reliant Medical Group, Worcester, Massachusetts
  - Ann Arbor VA Medical Center, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - HealthPartners Research Foundation, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
COPDGene phenotypic and genotypic data are available through dbGaP.

REFERENCES:
- [Derived] Zhang C, Konigsberg IR, He Y, Zhang J, Chikowore T, Feldman WB, Hu X, Ding Y, Pasaniuc B, Chang D, Chen Q, Lasky-Su JA, Hecker J, Tobin MD, Chen J, Kalra S, Pratte KA, Im HK, Wan ES, Manichaikul A, Silverman EK, Bowler RP, Lange LA, Ortega VE, Martin AR, Cho MH, Moll MR. Multi-Trait Polygenic Scores for COPD and COPD Exacerbations Implicate Druggable Proteins. medRxiv [Preprint]. 2025 Aug 26:2025.08.22.25334001. doi: 10.1101/2025.08.22.25334001. PMID 40909810
- [Derived] Awan HA, Chaudhary MFA, El-Sokkary AD, Hoffman EA, Comellas AP, Guo J, Barjaktarevic IZ, Barr RG, Bhatt SP, Bodduluri S, Bowler RP, Vargas Buonfiglio LG, Cooper CB, Fawzy A, Hastie AT, Labaki WW, Martinez FJ, Menchaca MG, O'Neal W, Paine R 3rd, Schroeder JD, Woodruff PG, Curtis JL, Reinhardt JM. Association of Lung Quantitative CT Scan Textures With Systemic Inflammation and Mortality in COPD. Chest. 2025 Nov;168(5):1107-1119. doi: 10.1016/j.chest.2025.04.017. Epub 2025 Apr 22. PMID 40268239
- [Derived] Kalra S, Hobbs B, Hunninghake GM, Menon AA, Putman R, Cutting C, Hatabu H, Silverman EK, Wan E, Cho MH, Moll M. The Association of Interstitial Lung Abnormalities and Preserved Ratio Impaired Spirometry With Mortality. Chest. 2025 Jul;168(1):136-145. doi: 10.1016/j.chest.2025.02.002. Epub 2025 Feb 11. PMID 39947315
- [Derived] Lee AN, Hsiao A, Hasenstab KA. Evaluating the Cumulative Benefit of Inspiratory CT, Expiratory CT, and Clinical Data for COPD Diagnosis and Staging through Deep Learning. Radiol Cardiothorac Imaging. 2024 Dec;6(6):e240005. doi: 10.1148/ryct.240005. PMID 39665633
- [Derived] van der Veer T, Andrinopoulou ER, Braunstahl GJ, Charbonnier JP, Kim V, Latisenko R, Lynch DA, Tiddens H. Association between automatic AI-based quantification of airway-occlusive mucus plugs and all-cause mortality in patients with COPD. Thorax. 2025 Jan 17;80(2):105-108. doi: 10.1136/thorax-2024-221928. PMID 39638548
- [Derived] Shirahata T, Enzer NA, Castro V, Chiles J, McDonald ML, Choi B, Diaz AA, Washko GR, San Jose Estepar R, Ash SY, Rahaghi FN. Effect of Common Medications on Longitudinal Pectoralis Muscle Area in Smokers. Chronic Obstr Pulm Dis. 2025 Jan 29;12(1):23-32. doi: 10.15326/jcopdf.2024.0557. PMID 39636057
- [Derived] Bell AJ, Ram S, Labaki WW, Murray S, Kazerooni EA, Galban S, Martinez FJ, Hatt CR, Wang JM, Ivanov V, McGettigan P, Khokhlovich E, Maiorino E, Suryadevara R, Boueiz A, Castaldi PJ, Mirkes EM, Zinovyev A, Gorban AN, Galban CJ, Han MK. Temporal Exploration of Chronic Obstructive Pulmonary Disease Phenotypes: Insights from the COPDGene and SPIROMICS Cohorts. Am J Respir Crit Care Med. 2025 Apr;211(4):569-576. doi: 10.1164/rccm.202401-0127OC. PMID 39269427
- [Derived] Yang HM, Ryu MH, Carey VJ, Young K, Kinney GL, Dransfield MT, Wade RC, Wells JM, Budoff MJ, Castaldi PJ, Hersh CP, Silverman EK. Differential Association of COPD Subtypes With Cardiovascular Events and COPD Exacerbations. Chest. 2024 Dec;166(6):1360-1370. doi: 10.1016/j.chest.2024.07.148. Epub 2024 Jul 31. PMID 39094733
- [Derived] Yang HM, Ryu MH, Carey VJ, Kinney GL, Hokanson JE, Dransfield MT, Hersh CP, Silverman EK; COPDGene Investigators dagger. Chronic Obstructive Pulmonary Disease Exacerbations Increase the Risk of Subsequent Cardiovascular Events: A Longitudinal Analysis of the COPDGene Study. J Am Heart Assoc. 2024 Jun 4;13(11):e033882. doi: 10.1161/JAHA.123.033882. Epub 2024 May 31. PMID 38818936
- [Derived] Nadeem SA, Comellas AP, Regan EA, Hoffman EA, Saha PK. Chest CT-based automated vertebral fracture assessment using artificial intelligence and morphologic features. Med Phys. 2024 Jun;51(6):4201-4218. doi: 10.1002/mp.17072. Epub 2024 May 9. PMID 38721977
- [Derived] Wang JM, Bell AJ, Ram S, Labaki WW, Hoff BA, Murray S, Kazerooni EA, Galban S, Hatt CR, Han MK, Galban CJ. Topologic Parametric Response Mapping Identifies Tissue Subtypes Associated with Emphysema Progression. Acad Radiol. 2024 Mar;31(3):1148-1159. doi: 10.1016/j.acra.2023.08.003. Epub 2023 Sep 2. PMID 37661554
- [Derived] Xie W, Jacobs C, Charbonnier JP, Slebos DJ, van Ginneken B. Emphysema subtyping on thoracic computed tomography scans using deep neural networks. Sci Rep. 2023 Aug 29;13(1):14147. doi: 10.1038/s41598-023-40116-6. PMID 37644032
- [Derived] Vestal BE, Ghosh D, Estepar RSJ, Kechris K, Fingerlin T, Carlson NE. Quantifying the spatial clustering characteristics of radiographic emphysema explains variability in pulmonary function. Sci Rep. 2023 Aug 24;13(1):13862. doi: 10.1038/s41598-023-40950-8. PMID 37620507
- [Derived] Amudala Puchakayala PR, Sthanam VL, Nakhmani A, Chaudhary MFA, Kizhakke Puliyakote A, Reinhardt JM, Zhang C, Bhatt SP, Bodduluri S. Radiomics for Improved Detection of Chronic Obstructive Pulmonary Disease in Low-Dose and Standard-Dose Chest CT Scans. Radiology. 2023 Jun;307(5):e222998. doi: 10.1148/radiol.222998. PMID 37338355
- [Derived] Hayden LP, Hobbs BD, Busch R, Cho MH, Liu M, Lopes-Ramos CM, Lomas DA, Bakke P, Gulsvik A, Silverman EK, Crapo JD, Beaty TH, Laird NM, Lange C, DeMeo DL. X chromosome associations with chronic obstructive pulmonary disease and related phenotypes: an X chromosome-wide association study. Respir Res. 2023 Feb 1;24(1):38. doi: 10.1186/s12931-023-02337-1. PMID 36726148
- [Derived] Gregory A, Xu Z, Pratte K, Lee S, Liu C, Chase R, Yun J, Saferali A, Hersh CP, Bowler R, Silverman E, Castaldi PJ, Boueiz A. Clustering-based COPD subtypes have distinct longitudinal outcomes and multi-omics biomarkers. BMJ Open Respir Res. 2022 Aug;9(1):e001182. doi: 10.1136/bmjresp-2021-001182. PMID 35999035
- [Derived] Balasubramanian A, Putcha N, MacIntyre NR, Jensen RL, Kinney G, Stringer WW, Hersh CP, Bowler RP, Casaburi R, Han MK, Porszasz J, Barr RG, Regan E, Make BJ, Hansel NN, Wise RA, McCormack MC. Diffusing Capacity and Mortality in Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2023 Jan;20(1):38-46. doi: 10.1513/AnnalsATS.202203-226OC. PMID 35969416
- [Derived] Oh AS, Baraghoshi D, Lynch DA, Ash SY, Crapo JD, Humphries SM; COPDGene Investigators. Emphysema Progression at CT by Deep Learning Predicts Functional Impairment and Mortality: Results from the COPDGene Study. Radiology. 2022 Sep;304(3):672-679. doi: 10.1148/radiol.213054. Epub 2022 May 17. PMID 35579519
- [Derived] Wan ES, Hokanson JE, Regan EA, Young KA, Make BJ, DeMeo DL, Mason SE, San Jose Estepar R, Crapo JD, Silverman EK. Significant Spirometric Transitions and Preserved Ratio Impaired Spirometry Among Ever Smokers. Chest. 2022 Mar;161(3):651-661. doi: 10.1016/j.chest.2021.09.021. Epub 2021 Sep 27. PMID 34592319
- [Derived] Yun JH, Lee C, Liu T, Liu S, Kim EY, Xu S, Curtis JL, Pinello L, Bowler RP, Silverman EK, Hersh CP, Zhou X. Hedgehog interacting protein-expressing lung fibroblasts suppress lymphocytic inflammation in mice. JCI Insight. 2021 Sep 8;6(17):e144575. doi: 10.1172/jci.insight.144575. PMID 34375314
- [Derived] Maselli DJ, Yen A, Wang W, Okajima Y, Dolliver WR, Mercugliano C, Anzueto A, Restrepo MI, Aksamit TR, Basavaraj A, Aliberti S, Young KA, Kinney GL, Wells JM, San Jose Estepar R, Lynch DA, Diaz AA. Small Airway Disease and Emphysema Are Associated with Future Exacerbations in Smokers with CT-derived Bronchiectasis and COPD: Results from the COPDGene Cohort. Radiology. 2021 Sep;300(3):706-714. doi: 10.1148/radiol.2021204052. Epub 2021 Jun 22. PMID 34156303
- [Derived] Tejwani V, Fawzy A, Putcha N, Castaldi PJ, Cho MH, Pratte KA, Bhatt SP, Lynch DA, Humphries SM, Kinney GL, D'Alessio FR, Hansel NN; COPDGene Investigators. Emphysema Progression and Lung Function Decline Among Angiotensin Converting Enzyme Inhibitors and Angiotensin-Receptor Blockade Users in the COPDGene Cohort. Chest. 2021 Oct;160(4):1245-1254. doi: 10.1016/j.chest.2021.05.007. Epub 2021 May 21. PMID 34029566
- [Derived] Luehrs RE, Moreau KL, Pierce GL, Wamboldt F, Aloia M, Weinberger HD, Make B, Bowler R, Crapo JD, Meschede K, Kozora E, Moser DJ, Hoth KF. Cognitive performance is lower among individuals with overlap syndrome than in individuals with COPD or obstructive sleep apnea alone: association with carotid artery stiffness. J Appl Physiol (1985). 2021 Jul 1;131(1):131-141. doi: 10.1152/japplphysiol.00477.2020. Epub 2021 May 13. PMID 33982592
- [Derived] Amaza IP, O'Shea AMJ, Fortis S, Comellas AP. Discordant Quantitative and Visual CT Assessments in the Diagnosis of Emphysema. Int J Chron Obstruct Pulmon Dis. 2021 May 3;16:1231-1242. doi: 10.2147/COPD.S284477. eCollection 2021. PMID 33976544
- [Derived] Wu TD, Fawzy A, Kinney GL, Bon J, Neupane M, Tejwani V, Hansel NN, Wise RA, Putcha N, McCormack MC. Metformin use and respiratory outcomes in asthma-COPD overlap. Respir Res. 2021 Feb 26;22(1):70. doi: 10.1186/s12931-021-01658-3. PMID 33637087
- [Derived] Pistenmaa CL, Nardelli P, Ash SY, Come CE, Diaz AA, Rahaghi FN, Barr RG, Young KA, Kinney GL, Simmons JP, Wade RC, Wells JM, Hokanson JE, Washko GR, San Jose Estepar R; COPDGene Investigators. Pulmonary Arterial Pruning and Longitudinal Change in Percent Emphysema and Lung Function: The Genetic Epidemiology of COPD Study. Chest. 2021 Aug;160(2):470-480. doi: 10.1016/j.chest.2021.01.084. Epub 2021 Feb 16. PMID 33607083
- [Derived] Ash SY, San Jose Estepar R, Fain SB, Tal-Singer R, Stockley RA, Nordenmark LH, Rennard S, Han MK, Merrill D, Humphries SM, Diaz AA, Mason SE, Rahaghi FN, Pistenmaa CL, Sciurba FC, Vegas-Sanchez-Ferrero G, Lynch DA, Washko GR; COPDGene Investigators and the COPD Biomarker Qualification Consortium. Relationship between Emphysema Progression at CT and Mortality in Ever-Smokers: Results from the COPDGene and ECLIPSE Cohorts. Radiology. 2021 Apr;299(1):222-231. doi: 10.1148/radiol.2021203531. Epub 2021 Feb 16. PMID 33591891
- [Derived] Moll M, Lutz SM, Ghosh AJ, Sakornsakolpat P, Hersh CP, Beaty TH, Dudbridge F, Tobin MD, Mittleman MA, Silverman EK, Hobbs BD, Cho MH. Relative contributions of family history and a polygenic risk score on COPD and related outcomes: COPDGene and ECLIPSE studies. BMJ Open Respir Res. 2020 Nov;7(1):e000755. doi: 10.1136/bmjresp-2020-000755. PMID 33239407
- [Derived] Billatos E, Ash SY, Duan F, Xu K, Romanoff J, Marques H, Moses E, Han MK, Regan EA, Bowler RP, Mason SE, Doyle TJ, San Jose Estepar R, Rosas IO, Ross JC, Xiao X, Liu H, Liu G, Sukumar G, Wilkerson M, Dalgard C, Stevenson C, Whitney D, Aberle D, Spira A, San Jose Estepar R, Lenburg ME, Washko GR; DECAMP and COPDGene Investigators. Distinguishing Smoking-Related Lung Disease Phenotypes Via Imaging and Molecular Features. Chest. 2021 Feb;159(2):549-563. doi: 10.1016/j.chest.2020.08.2115. Epub 2020 Sep 16. PMID 32946850
- [Derived] Baldomero AK, Wendt CH, Petersen A, Gaeckle NT, Han MK, Kunisaki KM; COPDGene Investigators. Impact of gastroesophageal reflux on longitudinal lung function and quantitative computed tomography in the COPDGene cohort. Respir Res. 2020 Aug 3;21(1):203. doi: 10.1186/s12931-020-01469-y. PMID 32746820
- [Derived] Bodduluri S, Nakhmani A, Reinhardt JM, Wilson CG, McDonald ML, Rudraraju R, Jaeger BC, Bhakta NR, Castaldi PJ, Sciurba FC, Zhang C, Bangalore PV, Bhatt SP. Deep neural network analyses of spirometry for structural phenotyping of chronic obstructive pulmonary disease. JCI Insight. 2020 Jul 9;5(13):e132781. doi: 10.1172/jci.insight.132781. PMID 32554922
- [Derived] Washko GR, Nardelli P, Ash SY, Rahaghi FN, Vegas Sanchez-Ferrero G, Come CE, Dransfield MT, Kalhan R, Han MK, Bhatt SP, Wells JM, Pistenmaa CL, Diaz AA, Ross JC, Rennard S, Querejeta Roca G, Shah AM, Young K, Kinney GL, Hokanson JE, Agusti A, San Jose Estepar R; COPDGene Investigators. Smaller Left Ventricle Size at Noncontrast CT Is Associated with Lower Mortality in COPDGene Participants. Radiology. 2020 Jul;296(1):208-215. doi: 10.1148/radiol.2020191793. Epub 2020 May 5. PMID 32368963
- [Derived] Hoth KF, Moreau KL, Weinberger HD, Holm KE, Meschede K, Crapo JD, Make BJ, Moser DJ, Kozora E, Bowler RP, Pierce GL, Ten Eyck P, Wamboldt FS. Carotid Artery Stiffness is Associated With Cognitive Performance in Former Smokers With and Without Chronic Obstructive Pulmonary Disease. J Am Heart Assoc. 2020 May 5;9(9):e014862. doi: 10.1161/JAHA.119.014862. Epub 2020 Apr 26. PMID 32338117
- [Derived] Lowe KE, Regan EA, Anzueto A, Austin E, Austin JHM, Beaty TH, Benos PV, Benway CJ, Bhatt SP, Bleecker ER, Bodduluri S, Bon J, Boriek AM, Boueiz AR, Bowler RP, Budoff M, Casaburi R, Castaldi PJ, Charbonnier JP, Cho MH, Comellas A, Conrad D, Costa Davis C, Criner GJ, Curran-Everett D, Curtis JL, DeMeo DL, Diaz AA, Dransfield MT, Dy JG, Fawzy A, Fleming M, Flenaugh EL, Foreman MG, Fortis S, Gebrekristos H, Grant S, Grenier PA, Gu T, Gupta A, Han MK, Hanania NA, Hansel NN, Hayden LP, Hersh CP, Hobbs BD, Hoffman EA, Hogg JC, Hokanson JE, Hoth KF, Hsiao A, Humphries S, Jacobs K, Jacobson FL, Kazerooni EA, Kim V, Kim WJ, Kinney GL, Koegler H, Lutz SM, Lynch DA, MacIntye NR Jr, Make BJ, Marchetti N, Martinez FJ, Maselli DJ, Mathews AM, McCormack MC, McDonald MN, McEvoy CE, Moll M, Molye SS, Murray S, Nath H, Newell JD Jr, Occhipinti M, Paoletti M, Parekh T, Pistolesi M, Pratte KA, Putcha N, Ragland M, Reinhardt JM, Rennard SI, Rosiello RA, Ross JC, Rossiter HB, Ruczinski I, San Jose Estepar R, Sciurba FC, Sieren JC, Singh H, Soler X, Steiner RM, Strand MJ, Stringer WW, Tal-Singer R, Thomashow B, Vegas Sanchez-Ferrero G, Walsh JW, Wan ES, Washko GR, Michael Wells J, Wendt CH, Westney G, Wilson A, Wise RA, Yen A, Young K, Yun J, Silverman EK, Crapo JD. COPDGene(R) 2019: Redefining the Diagnosis of Chronic Obstructive Pulmonary Disease. Chronic Obstr Pulm Dis. 2019 Nov;6(5):384-399. doi: 10.15326/jcopdf.6.5.2019.0149. PMID 31710793
- [Derived] Balasubramanian A, MacIntyre NR, Henderson RJ, Jensen RL, Kinney G, Stringer WW, Hersh CP, Bowler RP, Casaburi R, Han MK, Porszasz J, Barr RG, Make BJ, Wise RA, McCormack MC. Diffusing Capacity of Carbon Monoxide in Assessment of COPD. Chest. 2019 Dec;156(6):1111-1119. doi: 10.1016/j.chest.2019.06.035. Epub 2019 Jul 25. PMID 31352035
- [Derived] Kim W, Cho MH, Sakornsakolpat P, Lynch DA, Coxson HO, Tal-Singer R, Silverman EK, Beaty TH. DSP variants may be associated with longitudinal change in quantitative emphysema. Respir Res. 2019 Jul 19;20(1):160. doi: 10.1186/s12931-019-1097-8. PMID 31324189
- [Derived] Park J, Hobbs BD, Crapo JD, Make BJ, Regan EA, Humphries S, Carey VJ, Lynch DA, Silverman EK; COPDGene Investigators. Subtyping COPD by Using Visual and Quantitative CT Imaging Features. Chest. 2020 Jan;157(1):47-60. doi: 10.1016/j.chest.2019.06.015. Epub 2019 Jul 5. PMID 31283919
- [Derived] de la Hoz RE, Liu X, Celedon JC, Doucette JT, Jeon Y, Reeves AP, San Jose Estepar R. Association of Obesity with Quantitative Chest CT Measured Airway Wall Thickness in WTC Workers with Lower Airway Disease. Lung. 2019 Aug;197(4):517-522. doi: 10.1007/s00408-019-00246-z. Epub 2019 Jun 28. PMID 31254057
- [Derived] Harmouche R, Ash SY, Putman RK, Hunninghake GM, San Jose Estepar R, Martinez FJ, Choi AM, Lynch DA, Hatabu H, Han MK, Bowler RP, Kalhan R, Rosas IO, Washko GR, San Jose Estepar R; COPDGene Investigators. Objectively Measured Chronic Lung Injury on Chest CT. Chest. 2019 Dec;156(6):1149-1159. doi: 10.1016/j.chest.2019.05.020. Epub 2019 Jun 22. PMID 31233744
- [Derived] Maselli DJ, Bhatt SP, Anzueto A, Bowler RP, DeMeo DL, Diaz AA, Dransfield MT, Fawzy A, Foreman MG, Hanania NA, Hersh CP, Kim V, Kinney GL, Putcha N, Wan ES, Wells JM, Westney GE, Young KA, Silverman EK, Han MK, Make BJ. Clinical Epidemiology of COPD: Insights From 10 Years of the COPDGene Study. Chest. 2019 Aug;156(2):228-238. doi: 10.1016/j.chest.2019.04.135. Epub 2019 May 30. PMID 31154041
- [Derived] Kim V, Zhao H, Regan E, Han MK, Make BJ, Crapo JD, Jones PW, Curtis JL, Silverman EK, Criner GJ; COPDGene Investigators. The St. George's Respiratory Questionnaire Definition of Chronic Bronchitis May Be a Better Predictor of COPD Exacerbations Compared With the Classic Definition. Chest. 2019 Oct;156(4):685-695. doi: 10.1016/j.chest.2019.03.041. Epub 2019 May 15. PMID 31047955
- [Derived] Oudkerk SF, Mohamed Hoesein FAA, Oner FC, Verlaan JJ, de Jong PA, Kuperus JS, Cho M, McDonald ML, Lynch DA, Silverman EK, Crapo JD, Make BJ, Lowe KE, Regan EA. Diffuse Idiopathic Skeletal Hyperostosis in Smokers and Restrictive Spirometry Pattern: An Analysis of the COPDGene Cohort. J Rheumatol. 2020 Apr;47(4):531-538. doi: 10.3899/jrheum.181357. Epub 2019 May 1. PMID 31043539
- [Derived] Kuperus JS, Oudkerk SF, Foppen W, Mohamed Hoesein FA, Gielis WP, Waalwijk J, Regan EA, Lynch DA, Oner FC, de Jong PA, Verlaan JJ. Criteria for Early-Phase Diffuse Idiopathic Skeletal Hyperostosis: Development and Validation. Radiology. 2019 May;291(2):420-426. doi: 10.1148/radiol.2019181695. Epub 2019 Apr 2. PMID 30938626
- [Derived] Fortis S, Comellas A, Make BJ, Hersh CP, Bodduluri S, Georgopoulos D, Kim V, Criner GJ, Dransfield MT, Bhatt SP; COPDGene Investigators-Core Units: <italic>Administrative Center</italic>, COPDGene Investigators-Clinical Centers: <italic>Ann Arbor VA</italic>. Combined Forced Expiratory Volume in 1 Second and Forced Vital Capacity Bronchodilator Response, Exacerbations, and Mortality in Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2019 Jul;16(7):826-835. doi: 10.1513/AnnalsATS.201809-601OC. PMID 30908927
- [Derived] Bhatt SP, Bodduluri S, Raghav V, Bhakta NR, Wilson CG, Kim YI, Eberlein M, Sciurba FC, Han MK, Dransfield MT, Nakhmani A. The Peak Index: Spirometry Metric for Airflow Obstruction Severity and Heterogeneity. Ann Am Thorac Soc. 2019 Aug;16(8):982-989. doi: 10.1513/AnnalsATS.201811-812OC. PMID 30865842
- [Derived] Wan ES, Silverman EK. Reply to Marruchella: Preserved Ratio Impaired Spirometry and Interstitial Lung Abnormalities in Smokers. Am J Respir Crit Care Med. 2019 May 15;199(10):1293-1294. doi: 10.1164/rccm.201901-0018LE. No abstract available. PMID 30802417
- [Derived] Washko GR, Nardelli P, Ash SY, Vegas Sanchez-Ferrero G, Rahaghi FN, Come CE, Dransfield MT, Kalhan R, Han MK, Bhatt SP, Wells JM, Aaron CP, Diaz AA, Ross JC, Cuttica MJ, Labaki WW, Querejeta Roca G, Shah AM, Young K, Kinney GL, Hokanson JE, Agusti A, San Jose Estepar R. Arterial Vascular Pruning, Right Ventricular Size, and Clinical Outcomes in Chronic Obstructive Pulmonary Disease. A Longitudinal Observational Study. Am J Respir Crit Care Med. 2019 Aug 15;200(4):454-461. doi: 10.1164/rccm.201811-2063OC. PMID 30758975
- [Derived] Sakornsakolpat P, McCormack M, Bakke P, Gulsvik A, Make BJ, Crapo JD, Cho MH, Silverman EK. Genome-Wide Association Analysis of Single-Breath DlCO. Am J Respir Cell Mol Biol. 2019 May;60(5):523-531. doi: 10.1165/rcmb.2018-0384OC. PMID 30694715
- [Derived] Shaddox E, Peterson CB, Stingo FC, Hanania NA, Cruickshank-Quinn C, Kechris K, Bowler R, Vannucci M. Bayesian inference of networks across multiple sample groups and data types. Biostatistics. 2020 Jul 1;21(3):561-576. doi: 10.1093/biostatistics/kxy078. PMID 30590505
- [Derived] Miller ER, Putman RK, Diaz AA, Xu H, San Jose Estepar R, Araki T, Nishino M, Poli de Frias S, Hida T, Ross J, Coxson H, Dupuis J, O'Connor GT, Silverman EK, Rosas IO, Hatabu H, Washko G, Hunninghake GM. Increased Airway Wall Thickness in Interstitial Lung Abnormalities and Idiopathic Pulmonary Fibrosis. Ann Am Thorac Soc. 2019 Apr;16(4):447-454. doi: 10.1513/AnnalsATS.201806-424OC. PMID 30543456
- [Derived] Zhang C, Ramsey C, Berical A, Yu L, Leng L, McGinnis KA, Song Y, Michael H, McCormack MC, Allore H, Morris A, Crothers K, Bucala R, Lee PJ, Sauler M. A functional macrophage migration inhibitory factor promoter polymorphism is associated with reduced diffusing capacity. Am J Physiol Lung Cell Mol Physiol. 2019 Feb 1;316(2):L400-L405. doi: 10.1152/ajplung.00439.2018. Epub 2018 Dec 6. PMID 30520689
- [Derived] Wells JM, Parker MM, Oster RA, Bowler RP, Dransfield MT, Bhatt SP, Cho MH, Kim V, Curtis JL, Martinez FJ, Paine R 3rd, O'Neal W, Labaki WW, Kaner RJ, Barjaktarevic I, Han MK, Silverman EK, Crapo JD, Barr RG, Woodruff P, Castaldi PJ, Gaggar A; SPIROMICS and COPDGene Investigators. Elevated circulating MMP-9 is linked to increased COPD exacerbation risk in SPIROMICS and COPDGene. JCI Insight. 2018 Nov 15;3(22):e123614. doi: 10.1172/jci.insight.123614. PMID 30429371
- [Derived] Hayden LP, Cho MH, Raby BA, Beaty TH, Silverman EK, Hersh CP; COPDGene Investigators. Childhood asthma is associated with COPD and known asthma variants in COPDGene: a genome-wide association study. Respir Res. 2018 Oct 29;19(1):209. doi: 10.1186/s12931-018-0890-0. PMID 30373671
- [Derived] Boueiz A, Pham B, Chase R, Lamb A, Lee S, Naing ZZC, Cho MH, Parker MM, Sakornsakolpat P, Hersh CP, Crapo JD, Stergachis AB, Tal-Singer R, DeMeo DL, Silverman EK, Zhou X, Castaldi PJ; COPDGene investigators, by Core Units:, ECLIPSE Investigators:, GenKOLS Investigators:. Integrative Genomics Analysis Identifies ACVR1B as a Candidate Causal Gene of Emphysema Distribution. Am J Respir Cell Mol Biol. 2019 Apr;60(4):388-398. doi: 10.1165/rcmb.2018-0110OC. PMID 30335480
- [Derived] Bodduluri S, Puliyakote ASK, Gerard SE, Reinhardt JM, Hoffman EA, Newell JD Jr, Nath HP, Han MK, Washko GR, San Jose Estepar R, Dransfield MT, Bhatt SP; COPDGene Investigators. Airway fractal dimension predicts respiratory morbidity and mortality in COPD. J Clin Invest. 2018 Dec 3;128(12):5374-5382. doi: 10.1172/JCI120693. Epub 2018 Oct 29. PMID 30256767
- [Derived] Jiang Y, Chen S, McGuire D, Chen F, Liu M, Iacono WG, Hewitt JK, Hokanson JE, Krauter K, Laakso M, Li KW, Lutz SM, McGue M, Pandit A, Zajac GJM, Boehnke M, Abecasis GR, Vrieze SI, Zhan X, Jiang B, Liu DJ. Proper conditional analysis in the presence of missing data: Application to large scale meta-analysis of tobacco use phenotypes. PLoS Genet. 2018 Jul 17;14(7):e1007452. doi: 10.1371/journal.pgen.1007452. eCollection 2018 Jul. PMID 30016313
- [Derived] Prokopenko D, Sakornsakolpat P, Fier HL, Qiao D, Parker MM, McDonald MN, Manichaikul A, Rich SS, Barr RG, Williams CJ, Brantly ML, Lange C, Beaty TH, Crapo JD, Silverman EK, Cho MH. Whole-Genome Sequencing in Severe Chronic Obstructive Pulmonary Disease. Am J Respir Cell Mol Biol. 2018 Nov;59(5):614-622. doi: 10.1165/rcmb.2018-0088OC. PMID 29949718
- [Derived] Bhatt SP, Kazerooni EA, Newell JD Jr, Hokanson JE, Budoff MJ, Dass CA, Martinez CH, Bodduluri S, Jacobson FL, Yen A, Dransfield MT, Fuhrman C, Nath H; COPDGene Investigators. Visual Estimate of Coronary Artery Calcium Predicts Cardiovascular Disease in COPD. Chest. 2018 Sep;154(3):579-587. doi: 10.1016/j.chest.2018.05.037. Epub 2018 Jun 8. PMID 29890123
- [Derived] Wan ES, Fortis S, Regan EA, Hokanson J, Han MK, Casaburi R, Make BJ, Crapo JD, DeMeo DL, Silverman EK; COPDGene Investigators. Longitudinal Phenotypes and Mortality in Preserved Ratio Impaired Spirometry in the COPDGene Study. Am J Respir Crit Care Med. 2018 Dec 1;198(11):1397-1405. doi: 10.1164/rccm.201804-0663OC. PMID 29874098
- [Derived] Ash SY, Harmouche R, Ross JC, Diaz AA, Rahaghi FN, Vegas Sanchez-Ferrero G, Putman RK, Hunninghake GM, Onieva Onieva J, Martinez FJ, Choi AM, Bowler RP, Lynch DA, Hatabu H, Bhatt SP, Dransfield MT, Wells JM, Rosas IO, San Jose Estepar R, Washko GR; COPDGene Investigators. Interstitial Features at Chest CT Enhance the Deleterious Effects of Emphysema in the COPDGene Cohort. Radiology. 2018 Aug;288(2):600-609. doi: 10.1148/radiol.2018172688. Epub 2018 Jun 5. PMID 29869957
- [Derived] Diaz AA, Martinez CH, Harmouche R, Young TP, McDonald ML, Ross JC, Han ML, Bowler R, Make B, Regan EA, Silverman EK, Crapo J, Boriek AM, Kinney GL, Hokanson JE, Estepar RSJ, Washko GR. Pectoralis muscle area and mortality in smokers without airflow obstruction. Respir Res. 2018 Apr 10;19(1):62. doi: 10.1186/s12931-018-0771-6. PMID 29636050
- [Derived] Sakornsakolpat P, Morrow JD, Castaldi PJ, Hersh CP, Bosse Y, Silverman EK, Manichaikul A, Cho MH. Integrative genomics identifies new genes associated with severe COPD and emphysema. Respir Res. 2018 Mar 22;19(1):46. doi: 10.1186/s12931-018-0744-9. PMID 29566699
- [Derived] Ash SY, Harmouche R, Putman RK, Ross JC, Martinez FJ, Choi AM, Bowler RP, Regan EA, Curtis JL, Han MK, Boucher RC, O'Neal WK, Hatabu H, Lynch DA, Rosas IO, Hunninghake GM, San Jose Estepar R, Washko GR; COPDGene Investigators. Association between acute respiratory disease events and the MUC5B promoter polymorphism in smokers. Thorax. 2018 Nov;73(11):1071-1074. doi: 10.1136/thoraxjnl-2017-211208. Epub 2018 Feb 13. PMID 29440587
- [Derived] Fawzy A, Putcha N, Paulin LM, Aaron CP, Labaki WW, Han MK, Wise RA, Kanner RE, Bowler RP, Barr RG, Hansel NN; SPIROMICS and COPDGene Investigators. Association of thrombocytosis with COPD morbidity: the SPIROMICS and COPDGene cohorts. Respir Res. 2018 Jan 26;19(1):20. doi: 10.1186/s12931-018-0717-z. PMID 29373977
- [Derived] Morrow JD, Cho MH, Platig J, Zhou X, DeMeo DL, Qiu W, Celli B, Marchetti N, Criner GJ, Bueno R, Washko GR, Glass K, Quackenbush J, Silverman EK, Hersh CP. Ensemble genomic analysis in human lung tissue identifies novel genes for chronic obstructive pulmonary disease. Hum Genomics. 2018 Jan 15;12(1):1. doi: 10.1186/s40246-018-0132-z. PMID 29335020
- [Derived] Bhatt SP, Kim YI, Harrington KF, Hokanson JE, Lutz SM, Cho MH, DeMeo DL, Wells JM, Make BJ, Rennard SI, Washko GR, Foreman MG, Tashkin DP, Wise RA, Dransfield MT, Bailey WC; COPDGene Investigators. Smoking duration alone provides stronger risk estimates of chronic obstructive pulmonary disease than pack-years. Thorax. 2018 May;73(5):414-421. doi: 10.1136/thoraxjnl-2017-210722. Epub 2018 Jan 11. PMID 29326298
- [Derived] Hayden LP, Hardin ME, Qiu W, Lynch DA, Strand MJ, van Beek EJ, Crapo JD, Silverman EK, Hersh CP; COPDGene Investigators( *). Asthma Is a Risk Factor for Respiratory Exacerbations Without Increased Rate of Lung Function Decline: Five-Year Follow-up in Adult Smokers From the COPDGene Study. Chest. 2018 Feb;153(2):368-377. doi: 10.1016/j.chest.2017.11.038. Epub 2017 Dec 15. PMID 29248621
- [Derived] Halper-Stromberg E, Yun JH, Parker MM, Singer RT, Gaggar A, Silverman EK, Leach S, Bowler RP, Castaldi PJ. Systemic Markers of Adaptive and Innate Immunity Are Associated with Chronic Obstructive Pulmonary Disease Severity and Spirometric Disease Progression. Am J Respir Cell Mol Biol. 2018 Apr;58(4):500-509. doi: 10.1165/rcmb.2017-0373OC. PMID 29206476
- [Derived] Diaz AA, Strand M, Coxson HO, Ross JC, San Jose Estepar R, Lynch D, van Rikxoort EM, Rosas IO, Hunninghake GM, Putman RK, Hatabu H, Yen A, Kinney GL, Hokanson JE, Silverman EK, Crapo J, Washko GR. Disease Severity Dependence of the Longitudinal Association Between CT Lung Density and Lung Function in Smokers. Chest. 2018 Mar;153(3):638-645. doi: 10.1016/j.chest.2017.10.012. Epub 2017 Oct 21. PMID 29066389
- [Derived] Boueiz A, Chang Y, Cho MH, Washko GR, San Jose Estepar R, Bowler RP, Crapo JD, DeMeo DL, Dy JG, Silverman EK, Castaldi PJ; COPDGene Investigators. Lobar Emphysema Distribution Is Associated With 5-Year Radiological Disease Progression. Chest. 2018 Jan;153(1):65-76. doi: 10.1016/j.chest.2017.09.022. Epub 2017 Sep 21. PMID 28943279
- [Derived] Brunette AM, Holm KE, Wamboldt FS, Kozora E, Moser DJ, Make BJ, Crapo JD, Meschede K, Weinberger HD, Moreau KL, Bowler RP, Hoth KF. Subjective cognitive complaints and neuropsychological performance in former smokers with and without chronic obstructive pulmonary disease. J Clin Exp Neuropsychol. 2018 May;40(4):411-422. doi: 10.1080/13803395.2017.1356912. Epub 2017 Aug 2. PMID 28766459
- [Derived] Bodduluri S, Reinhardt JM, Hoffman EA, Newell JD Jr, Nath H, Dransfield MT, Bhatt SP; COPDGene Investigators. Signs of Gas Trapping in Normal Lung Density Regions in Smokers. Am J Respir Crit Care Med. 2017 Dec 1;196(11):1404-1410. doi: 10.1164/rccm.201705-0855OC. PMID 28707983
- [Derived] Bhatt SP, Bodduluri S, Hoffman EA, Newell JD Jr, Sieren JC, Dransfield MT, Reinhardt JM; COPDGene Investigators. Computed Tomography Measure of Lung at Risk and Lung Function Decline in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2017 Sep 1;196(5):569-576. doi: 10.1164/rccm.201701-0050OC. PMID 28481639
- [Derived] Bhatt SP, Vegas-Sanchez-Ferrero G, Rahaghi FN, MacLean ES, Gonzalez-Serrano G, Come CE, Kinney GL, Hokanson JE, Budoff MJ, Cuttica MJ, Wells JM, Estepar RSJ, Washko GR. Cardiac Morphometry on Computed Tomography and Exacerbation Reduction with beta-Blocker Therapy in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2017 Dec 1;196(11):1484-1488. doi: 10.1164/rccm.201702-0399LE. No abstract available. PMID 28441027
- [Derived] Hodgson S, Griffin TJ, Reilly C, Harvey S, Witthuhn BA, Sandri BJ, Kunisaki KM, Wendt CH. Plasma sphingolipids in HIV-associated chronic obstructive pulmonary disease. BMJ Open Respir Res. 2017 Apr 3;4(1):e000180. doi: 10.1136/bmjresp-2017-000180. eCollection 2017. PMID 28409005
- [Derived] Martinez CH, Freeman CM, Nelson JD, Murray S, Wang X, Budoff MJ, Dransfield MT, Hokanson JE, Kazerooni EA, Kinney GL, Regan EA, Wells JM, Martinez FJ, Han MK, Curtis JL; COPDGene Investigators. GDF-15 plasma levels in chronic obstructive pulmonary disease are associated with subclinical coronary artery disease. Respir Res. 2017 Feb 28;18(1):42. doi: 10.1186/s12931-017-0521-1. PMID 28245821
- [Derived] Bodduluri S, Bhatt SP, Hoffman EA, Newell JD Jr, Martinez CH, Dransfield MT, Han MK, Reinhardt JM; COPDGene Investigators. Biomechanical CT metrics are associated with patient outcomes in COPD. Thorax. 2017 May;72(5):409-414. doi: 10.1136/thoraxjnl-2016-209544. Epub 2017 Jan 2. PMID 28044005
- [Derived] Wells JM, Estepar RS, McDonald MN, Bhatt SP, Diaz AA, Bailey WC, Jacobson FL, Dransfield MT, Washko GR, Make BJ, Casaburi R, van Beek EJ, Hoffman EA, Sciurba FC, Crapo JD, Silverman EK, Hersh CP; COPDGene Investigators. Clinical, physiologic, and radiographic factors contributing to development of hypoxemia in moderate to severe COPD: a cohort study. BMC Pulm Med. 2016 Dec 1;16(1):169. doi: 10.1186/s12890-016-0331-0. PMID 27903260
- [Derived] Diaz AA, Young TP, Maselli DJ, Martinez CH, Gill R, Nardelli P, Wang W, Kinney GL, Hokanson JE, Washko GR, San Jose Estepar R. Quantitative CT Measures of Bronchiectasis in Smokers. Chest. 2017 Jun;151(6):1255-1262. doi: 10.1016/j.chest.2016.11.024. Epub 2016 Nov 24. PMID 27890712
- [Derived] Boueiz A, Lutz SM, Cho MH, Hersh CP, Bowler RP, Washko GR, Halper-Stromberg E, Bakke P, Gulsvik A, Laird NM, Beaty TH, Coxson HO, Crapo JD, Silverman EK, Castaldi PJ, DeMeo DL; COPDGene and ECLIPSE Investigators. Genome-Wide Association Study of the Genetic Determinants of Emphysema Distribution. Am J Respir Crit Care Med. 2017 Mar 15;195(6):757-771. doi: 10.1164/rccm.201605-0997OC. PMID 27669027
- [Derived] Dransfield MT, Kunisaki KM, Strand MJ, Anzueto A, Bhatt SP, Bowler RP, Criner GJ, Curtis JL, Hanania NA, Nath H, Putcha N, Roark SE, Wan ES, Washko GR, Wells JM, Wendt CH, Make BJ; COPDGene Investigators. Acute Exacerbations and Lung Function Loss in Smokers with and without Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2017 Feb 1;195(3):324-330. doi: 10.1164/rccm.201605-1014OC. PMID 27556408
- [Derived] Diaz AA, Young TP, Maselli DJ, Martinez CH, Maclean ES, Yen A, Dass C, Simpson SA, Lynch DA, Kinney GL, Hokanson JE, Washko GR, San Jose Estepar R. Bronchoarterial ratio in never-smokers adults: Implications for bronchial dilation definition. Respirology. 2017 Jan;22(1):108-113. doi: 10.1111/resp.12875. Epub 2016 Aug 18. PMID 27538197
- [Derived] Hayden LP, Cho MH, McDonald MN, Crapo JD, Beaty TH, Silverman EK, Hersh CP; COPDGene Investigators *. Susceptibility to Childhood Pneumonia: A Genome-Wide Analysis. Am J Respir Cell Mol Biol. 2017 Jan;56(1):20-28. doi: 10.1165/rcmb.2016-0101OC. PMID 27508494
- [Derived] Bhatt SP, Bodduluri S, Newell JD, Hoffman EA, Sieren JC, Han MK, Dransfield MT, Reinhardt JM; COPDGene Investigators. CT-derived Biomechanical Metrics Improve Agreement Between Spirometry and Emphysema. Acad Radiol. 2016 Oct;23(10):1255-63. doi: 10.1016/j.acra.2016.02.002. Epub 2016 Apr 4. PMID 27055745
- [Derived] Busch R, Han MK, Bowler RP, Dransfield MT, Wells JM, Regan EA, Hersh CP; COPDGene Investigators. Risk factors for COPD exacerbations in inhaled medication users: the COPDGene study biannual longitudinal follow-up prospective cohort. BMC Pulm Med. 2016 Feb 10;16:28. doi: 10.1186/s12890-016-0191-7. PMID 26861867
- [Derived] Martinez CH, Diaz AA, Parulekar AD, Rennard SI, Kanner RE, Hansel NN, Couper D, Holm KE, Hoth KF, Curtis JL, Martinez FJ, Hanania NA, Regan EA, Paine R 3rd, Cigolle CT, Han MK; COPDGene and SPIROMICS Investigators. Age-Related Differences in Health-Related Quality of Life in COPD: An Analysis of the COPDGene and SPIROMICS Cohorts. Chest. 2016 Apr;149(4):927-35. doi: 10.1016/j.chest.2015.11.025. Epub 2015 Dec 17. PMID 26836895
- [Derived] Bhatt SP, Soler X, Wang X, Murray S, Anzueto AR, Beaty TH, Boriek AM, Casaburi R, Criner GJ, Diaz AA, Dransfield MT, Curran-Everett D, Galban CJ, Hoffman EA, Hogg JC, Kazerooni EA, Kim V, Kinney GL, Lagstein A, Lynch DA, Make BJ, Martinez FJ, Ramsdell JW, Reddy R, Ross BD, Rossiter HB, Steiner RM, Strand MJ, van Beek EJ, Wan ES, Washko GR, Wells JM, Wendt CH, Wise RA, Silverman EK, Crapo JD, Bowler RP, Han MK; COPDGene Investigators. Association between Functional Small Airway Disease and FEV1 Decline in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2016 Jul 15;194(2):178-84. doi: 10.1164/rccm.201511-2219OC. PMID 26808615
- [Derived] Hobbs BD, Parker MM, Chen H, Lao T, Hardin M, Qiao D, Hawrylkiewicz I, Sliwinski P, Yim JJ, Kim WJ, Kim DK, Castaldi PJ, Hersh CP, Morrow J, Celli BR, Pinto-Plata VM, Criner GJ, Marchetti N, Bueno R, Agusti A, Make BJ, Crapo JD, Calverley PM, Donner CF, Lomas DA, Wouters EF, Vestbo J, Pare PD, Levy RD, Rennard SI, Zhou X, Laird NM, Lin X, Beaty TH, Silverman EK, Cho MH; NETT Genetics Investigators; ECLIPSE Investigators; COPDGene Investigators; International COPD Genetics Network Investigators. Exome Array Analysis Identifies a Common Variant in IL27 Associated with Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2016 Jul 1;194(1):48-57. doi: 10.1164/rccm.201510-2053OC. PMID 26771213
- [Derived] Qiao D, Lange C, Beaty TH, Crapo JD, Barnes KC, Bamshad M, Hersh CP, Morrow J, Pinto-Plata VM, Marchetti N, Bueno R, Celli BR, Criner GJ, Silverman EK, Cho MH; Lung GO; NHLBI Exome Sequencing Project; COPDGene Investigators. Exome Sequencing Analysis in Severe, Early-Onset Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2016 Jun 15;193(12):1353-63. doi: 10.1164/rccm.201506-1223OC. PMID 26736064
- [Derived] Lutz SM, Cho MH, Young K, Hersh CP, Castaldi PJ, McDonald ML, Regan E, Mattheisen M, DeMeo DL, Parker M, Foreman M, Make BJ, Jensen RL, Casaburi R, Lomas DA, Bhatt SP, Bakke P, Gulsvik A, Crapo JD, Beaty TH, Laird NM, Lange C, Hokanson JE, Silverman EK; ECLIPSE Investigators; COPDGene Investigators. A genome-wide association study identifies risk loci for spirometric measures among smokers of European and African ancestry. BMC Genet. 2015 Dec 3;16:138. doi: 10.1186/s12863-015-0299-4. PMID 26634245
- [Derived] Hayden LP, Hobbs BD, Cohen RT, Wise RA, Checkley W, Crapo JD, Hersh CP; COPDGene Investigators. Childhood pneumonia increases risk for chronic obstructive pulmonary disease: the COPDGene study. Respir Res. 2015 Sep 21;16(1):115. doi: 10.1186/s12931-015-0273-8. PMID 26392057
- [Derived] Bhatt SP, Wells JM, Kinney GL, Washko GR Jr, Budoff M, Kim YI, Bailey WC, Nath H, Hokanson JE, Silverman EK, Crapo J, Dransfield MT; COPDGene Investigators. beta-Blockers are associated with a reduction in COPD exacerbations. Thorax. 2016 Jan;71(1):8-14. doi: 10.1136/thoraxjnl-2015-207251. Epub 2015 Aug 17. PMID 26283710
- [Derived] Batmanghelich NK, Saeedi A, Cho M, Estepar RS, Golland P. Generative Method to Discover Genetically Driven Image Biomarkers. Inf Process Med Imaging. 2015;24:30-42. doi: 10.1007/978-3-319-19992-4_3. PMID 26221665
- [Derived] Cho MH, Castaldi PJ, Hersh CP, Hobbs BD, Barr RG, Tal-Singer R, Bakke P, Gulsvik A, San Jose Estepar R, Van Beek EJ, Coxson HO, Lynch DA, Washko GR, Laird NM, Crapo JD, Beaty TH, Silverman EK; NETT Genetics, ECLIPSE, and COPDGene Investigators. A Genome-Wide Association Study of Emphysema and Airway Quantitative Imaging Phenotypes. Am J Respir Crit Care Med. 2015 Sep 1;192(5):559-69. doi: 10.1164/rccm.201501-0148OC. PMID 26030696
- [Derived] Wells JM, Iyer AS, Rahaghi FN, Bhatt SP, Gupta H, Denney TS, Lloyd SG, Dell'Italia LJ, Nath H, Estepar RS, Washko GR, Dransfield MT. Pulmonary artery enlargement is associated with right ventricular dysfunction and loss of blood volume in small pulmonary vessels in chronic obstructive pulmonary disease. Circ Cardiovasc Imaging. 2015 Apr;8(4):10.1161/CIRCIMAGING.114.002546 e002546. doi: 10.1161/CIRCIMAGING.114.002546. PMID 25855668
- [Derived] Hersh CP, Make BJ, Lynch DA, Barr RG, Bowler RP, Calverley PM, Castaldi PJ, Cho MH, Coxson HO, DeMeo DL, Foreman MG, Han MK, Harshfield BJ, Hokanson JE, Lutz S, Ramsdell JW, Regan EA, Rennard SI, Schroeder JD, Sciurba FC, Steiner RM, Tal-Singer R, van Beek E Jr, Silverman EK, Crapo JD; COPDGene and ECLIPSE Investigators. Non-emphysematous chronic obstructive pulmonary disease is associated with diabetes mellitus. BMC Pulm Med. 2014 Oct 24;14:164. doi: 10.1186/1471-2466-14-164. PMID 25341556
- [Derived] Diaz AA, Hardin ME, Come CE, San Jose Estepar R, Ross JC, Kurugol S, Okajima Y, Han MK, Kim V, Ramsdell J, Silverman EK, Crapo JD, Lynch DA, Make B, Barr RG, Hersh CP, Washko GR; COPDGene Investigators. Childhood-onset asthma in smokers. association between CT measures of airway size, lung function, and chronic airflow obstruction. Ann Am Thorac Soc. 2014 Nov;11(9):1371-8. doi: 10.1513/AnnalsATS.201403-095OC. PMID 25296268
- [Derived] Hobbs BD, Foreman MG, Bowler R, Jacobson F, Make BJ, Castaldi PJ, San Jose Estepar R, Silverman EK, Hersh CP; COPDGene Investigators. Pneumothorax risk factors in smokers with and without chronic obstructive pulmonary disease. Ann Am Thorac Soc. 2014 Nov;11(9):1387-94. doi: 10.1513/AnnalsATS.201405-224OC. PMID 25295410
- [Derived] Lee JH, Cho MH, Hersh CP, McDonald ML, Crapo JD, Bakke PS, Gulsvik A, Comellas AP, Wendt CH, Lomas DA, Kim V, Silverman EK; COPDGene and ECLIPSE Investigators. Genetic susceptibility for chronic bronchitis in chronic obstructive pulmonary disease. Respir Res. 2014 Sep 21;15(1):113. doi: 10.1186/s12931-014-0113-2. PMID 25241909
- [Derived] Lee JH, McDonald ML, Cho MH, Wan ES, Castaldi PJ, Hunninghake GM, Marchetti N, Lynch DA, Crapo JD, Lomas DA, Coxson HO, Bakke PS, Silverman EK, Hersh CP; COPDGene and ECLIPSE Investigators. DNAH5 is associated with total lung capacity in chronic obstructive pulmonary disease. Respir Res. 2014 Aug 20;15(1):97. doi: 10.1186/s12931-014-0097-y. PMID 25134640
- [Derived] Wan ES, Castaldi PJ, Cho MH, Hokanson JE, Regan EA, Make BJ, Beaty TH, Han MK, Curtis JL, Curran-Everett D, Lynch DA, DeMeo DL, Crapo JD, Silverman EK; COPDGene Investigators. Epidemiology, genetics, and subtyping of preserved ratio impaired spirometry (PRISm) in COPDGene. Respir Res. 2014 Aug 6;15(1):89. doi: 10.1186/s12931-014-0089-y. PMID 25096860
- [Derived] Bhatt SP, Sieren JC, Newell JD Jr, Comellas AP, Hoffman EA. Disproportionate contribution of right middle lobe to emphysema and gas trapping on computed tomography. PLoS One. 2014 Jul 23;9(7):e102807. doi: 10.1371/journal.pone.0102807. eCollection 2014. PMID 25054539
- [Derived] Castaldi PJ, Cho MH, San Jose Estepar R, McDonald ML, Laird N, Beaty TH, Washko G, Crapo JD, Silverman EK; COPDGene Investigators. Genome-wide association identifies regulatory Loci associated with distinct local histogram emphysema patterns. Am J Respir Crit Care Med. 2014 Aug 15;190(4):399-409. doi: 10.1164/rccm.201403-0569OC. PMID 25006744
- [Derived] McDonald ML, Cho MH, Sorheim IC, Lutz SM, Castaldi PJ, Lomas DA, Coxson HO, Edwards LD, MacNee W, Vestbo J, Yates JC, Agusti A, Calverley PM, Celli B, Crim C, Rennard SI, Wouters EF, Bakke P, Tal-Singer R, Miller BE, Gulsvik A, Casaburi R, Wells JM, Regan EA, Make BJ, Hokanson JE, Lange C, Crapo JD, Beaty TH, Silverman EK, Hersh CP; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints and COPDGene Investigators. Common genetic variants associated with resting oxygenation in chronic obstructive pulmonary disease. Am J Respir Cell Mol Biol. 2014 Nov;51(5):678-87. doi: 10.1165/rcmb.2014-0135OC. PMID 24825563
- [Derived] Manichaikul A, Hoffman EA, Smolonska J, Gao W, Cho MH, Baumhauer H, Budoff M, Austin JH, Washko GR, Carr JJ, Kaufman JD, Pottinger T, Powell CA, Wijmenga C, Zanen P, Groen HJ, Postma DS, Wanner A, Rouhani FN, Brantly ML, Powell R, Smith BM, Rabinowitz D, Raffel LJ, Hinckley Stukovsky KD, Crapo JD, Beaty TH, Hokanson JE, Silverman EK, Dupuis J, O'Connor GT, Boezen HM, Rich SS, Barr RG. Genome-wide study of percent emphysema on computed tomography in the general population. The Multi-Ethnic Study of Atherosclerosis Lung/SNP Health Association Resource Study. Am J Respir Crit Care Med. 2014 Feb 15;189(4):408-18. doi: 10.1164/rccm.201306-1061OC. PMID 24383474
- [Derived] Han MK, Muellerova H, Curran-Everett D, Dransfield MT, Washko GR, Regan EA, Bowler RP, Beaty TH, Hokanson JE, Lynch DA, Jones PW, Anzueto A, Martinez FJ, Crapo JD, Silverman EK, Make BJ. GOLD 2011 disease severity classification in COPDGene: a prospective cohort study. Lancet Respir Med. 2013 Mar;1(1):43-50. doi: 10.1016/S2213-2600(12)70044-9. Epub 2012 Sep 3. PMID 24321803
- [Derived] Martinez CH, Kim V, Chen Y, Kazerooni EA, Murray S, Criner GJ, Curtis JL, Regan EA, Wan E, Hersh CP, Silverman EK, Crapo JD, Martinez FJ, Han MK; COPDGene Investigators. The clinical impact of non-obstructive chronic bronchitis in current and former smokers. Respir Med. 2014 Mar;108(3):491-9. doi: 10.1016/j.rmed.2013.11.003. Epub 2013 Nov 15. PMID 24280543
- [Derived] Diaz AA, Han MK, Come CE, San Jose Estepar R, Ross JC, Kim V, Dransfield MT, Curran-Everett D, Schroeder JD, Lynch DA, Tschirren J, Silverman EK, Washko GR. Effect of emphysema on CT scan measures of airway dimensions in smokers. Chest. 2013 Mar;143(3):687-693. doi: 10.1378/chest.12-0039. PMID 23460155
- [Derived] Wells JM, Washko GR, Han MK, Abbas N, Nath H, Mamary AJ, Regan E, Bailey WC, Martinez FJ, Westfall E, Beaty TH, Curran-Everett D, Curtis JL, Hokanson JE, Lynch DA, Make BJ, Crapo JD, Silverman EK, Bowler RP, Dransfield MT; COPDGene Investigators; ECLIPSE Study Investigators. Pulmonary arterial enlargement and acute exacerbations of COPD. N Engl J Med. 2012 Sep 6;367(10):913-21. doi: 10.1056/NEJMoa1203830. Epub 2012 Sep 3. PMID 22938715
- [Derived] Doyle TJ, Washko GR, Fernandez IE, Nishino M, Okajima Y, Yamashiro T, Divo MJ, Celli BR, Sciurba FC, Silverman EK, Hatabu H, Rosas IO, Hunninghake GM; COPDGene Investigators. Interstitial lung abnormalities and reduced exercise capacity. Am J Respir Crit Care Med. 2012 Apr 1;185(7):756-62. doi: 10.1164/rccm.201109-1618OC. Epub 2012 Jan 20. PMID 22268134
- [Derived] Xu JF, Washko GR, Nakahira K, Hatabu H, Patel AS, Fernandez IE, Nishino M, Okajima Y, Yamashiro T, Ross JC, Estepar RS, Diaz AA, Li HP, Qu JM, Himes BE, Come CE, D'Aco K, Martinez FJ, Han MK, Lynch DA, Crapo JD, Morse D, Ryter SW, Silverman EK, Rosas IO, Choi AM, Hunninghake GM; COPDGene Investigators. Statins and pulmonary fibrosis: the potential role of NLRP3 inflammasome activation. Am J Respir Crit Care Med. 2012 Mar 1;185(5):547-56. doi: 10.1164/rccm.201108-1574OC. Epub 2012 Jan 12. PMID 22246178
- [Derived] Hardin M, Silverman EK, Barr RG, Hansel NN, Schroeder JD, Make BJ, Crapo JD, Hersh CP; COPDGene Investigators. The clinical features of the overlap between COPD and asthma. Respir Res. 2011 Sep 27;12(1):127. doi: 10.1186/1465-9921-12-127. PMID 21951550
- [Derived] Diaz AA, Come CE, Ross JC, San Jose Estepar R, Han MK, Loring SH, Silverman EK, Washko GR; COPDGene Investigators. Association between airway caliber changes with lung inflation and emphysema assessed by volumetric CT scan in subjects with COPD. Chest. 2012 Mar;141(3):736-744. doi: 10.1378/chest.11-1026. Epub 2011 Sep 22. PMID 21940776
- [Derived] Han MK, Curran-Everett D, Dransfield MT, Criner GJ, Zhang L, Murphy JR, Hansel NN, DeMeo DL, Hanania NA, Regan EA, Make BJ, Martinez FJ, Westney GE, Foreman MG; COPDGene Investigators. Racial differences in quality of life in patients with COPD. Chest. 2011 Nov;140(5):1169-1176. doi: 10.1378/chest.10-2869. Epub 2011 Jun 2. PMID 21636665
- [Derived] Wan ES, Hokanson JE, Murphy JR, Regan EA, Make BJ, Lynch DA, Crapo JD, Silverman EK; COPDGene Investigators. Clinical and radiographic predictors of GOLD-unclassified smokers in the COPDGene study. Am J Respir Crit Care Med. 2011 Jul 1;184(1):57-63. doi: 10.1164/rccm.201101-0021OC. Epub 2011 Apr 14. PMID 21493737
- [Derived] Kim V, Han MK, Vance GB, Make BJ, Newell JD, Hokanson JE, Hersh CP, Stinson D, Silverman EK, Criner GJ; COPDGene Investigators. The chronic bronchitic phenotype of COPD: an analysis of the COPDGene Study. Chest. 2011 Sep;140(3):626-633. doi: 10.1378/chest.10-2948. Epub 2011 Apr 7. PMID 21474571
- [Derived] Kim DK, Jacobson FL, Washko GR, Casaburi R, Make BJ, Crapo JD, Silverman EK, Hersh CP. Clinical and radiographic correlates of hypoxemia and oxygen therapy in the COPDGene study. Respir Med. 2011 Aug;105(8):1211-21. doi: 10.1016/j.rmed.2011.02.015. Epub 2011 Mar 10. PMID 21396809
- [Derived] Washko GR, Hunninghake GM, Fernandez IE, Nishino M, Okajima Y, Yamashiro T, Ross JC, Estepar RS, Lynch DA, Brehm JM, Andriole KP, Diaz AA, Khorasani R, D'Aco K, Sciurba FC, Silverman EK, Hatabu H, Rosas IO; COPDGene Investigators. Lung volumes and emphysema in smokers with interstitial lung abnormalities. N Engl J Med. 2011 Mar 10;364(10):897-906. doi: 10.1056/NEJMoa1007285. PMID 21388308
- [Derived] Kim DK, Hersh CP, Washko GR, Hokanson JE, Lynch DA, Newell JD, Murphy JR, Crapo JD, Silverman EK; COPD Gene Investigators. Epidemiology, radiology, and genetics of nicotine dependence in COPD. Respir Res. 2011 Jan 13;12(1):9. doi: 10.1186/1465-9921-12-9. PMID 21232152